CLINICAL TRIAL: NCT04872491
Title: A Prospective, Multicenter, Single-arm, Observational Study to Evaluate the Safety and Effectiveness of Vedolizumab in Real-World Clinical Practice in China
Brief Title: A Study of Vedolizumab in Adults in Real-World Practice
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5064
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With UC or CD: Participants diagnosed with UC or CD who are prescribed and will start treatment with vedolizumab 300 milligram (mg), infusion, intravenously, at Weeks 0, 2, 6, and every 8 weeks thereafter for up to 54 weeks will be observed prospectively for 72 weeks.

SUMMARY:
Vedolizumab is a medicine that is currently prescribed for adults with moderately to severely active ulcerative colitis or Crohn's disease.

In this study, adults with ulcerative colitis or Crohn's disease will be treated with vedolizumab according to their clinic's standard practice. The main aim of the study is to check if participants have side effects from vedolizumab.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with UC or CD who are prescribed and will start vedolizumab in the real word setting for the first time.

This study will evaluate the safety and effectiveness of vedolizumab in a routine clinical practice setting under real world conditions.

The study will enroll approximately 500 participants. The data will be prospectively collected, at the centers from routinely scheduled follow-up visits and recorded into electronic data capture (eDC). All participants will be enrolled in a single observational group:

• Participants with UC or CD

This multi-center trial will be conducted in China. The overall duration of the study will be approximately 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with UC or CD
2. Firstly prescribed with vedolizumab

Exclusion Criteria:

1. Currently enrolled in or plan to participate in any other clinical trials (that is, interventional study)
2. Contraindicated for vedolizumab according to product package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with UC or CD, who have been prescribed and will start vedolizumab in clinical practice will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to Week 72
Percentage of Participants With Serious Adverse Events (SAEs) | Up to Week 72
Percentage of Participants With Adverse Events of Special Interests (AESIs) | Up to Week 72
Percentage of Participants With Adverse Drug Reactions (ADRs) | Up to Week 72

SECONDARY OUTCOMES:
Percentage of Participants With Ulcerative Colitis (UC) Achieving Clinical Response Based on Partial Mayo Score | Week 14
  Clinical response in UC is defined as greater than or equal to (>=) 2 points reduction in partial mayo clinic score and >=25 percent (%) decrease from baseline score accompanied with >=1 point decrease in rectal bleeding sub-score or absolute rectal bleeding sub-score less than or equal to (<=) 1 point. Partial mayo score is an instrument designed to measure disease activity of UC. It consists of 3 sub-scores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease.
Percentage of Participants With Crohn's Disease (CD) Achieving Clinical Response Based on Harvey-Bradshaw Index (HBI) | Week 14
  Clinical response in CD is defined as >=3-point decrease in the HBI score. HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0 equal to [=] very well to 4 = terrible), abdominal pain (0 = none to 3 = severe), number of liquid or soft stools per day, abdominal mass (0 = none to 3 = definite and tender), and complications (8 items; 1 score per item). The total score is sum of sub-scores, where score less than (<) 5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and greater than (>) 16 = severe disease activity.
Percentage of Participants With UC Achieving Clinical Remission Based on Partial Mayo Score | Week 54
  Clinical remission in UC is defined as partial mayo clinic score <=2 with no sub-score >1. Partial mayo score is an instrument designed to measure disease activity of UC. It consists of 3 sub-scores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease.
Percentage of Participants With CD Achieving Clinical Remission Based on HBI | Week 54
  Clinical remission in CD is defined as HBI score of <=4 points. HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0 = very well to 4 = terrible), abdominal pain (0 = none to 3 = severe), number of liquid or soft stools per day, abdominal mass (0 = none to 3 = definite and tender), and complications (8 items; 1 score per item). The total score is sum of sub-scores, where score <5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and >16 = severe disease activity.
Percentage of Participants With UC Achieving Endoscopic Remission | Week 54
  Endoscopic remission in UC is defined as mayo endoscopic sub-score <=1. Mayo endoscopic sub-score (findings on endoscopy), each graded from 0 to 3 where 0 = Normal mucosa or inactive disease, 1 = Mild activity (erythema, decreased vascular pattern, mild friability), 2 = Moderate activity (marked erythema, lack of vascular pattern, friability, erosions), 3 = Severe activity (spontaneous bleeding, large ulcerations). Higher scores indicating more severe disease.
Percentage of Participants With CD Achieving Endoscopic Remission | Week 54
  Endoscopic remission in CD is defined as absence of any ulcers excluding aphthous ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (40):
- China (40):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Heilongjiang Provincial Hospital (Nanshang ), Harbin, Heilongjiang
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - The Third Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital Original Region, Suzhou, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The 2nd Hospital of XiAn Jiaotong University, Xi'an, Shan'xi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/6093e1a3ef0b71001e743c46